CLINICAL TRIAL: NCT03104036
Title: Faecal Bacteriotherapy for Ulcerative Colitis
Acronym: FACTU
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Collaborators: Institute of Animal Physiology and Genetics Academy of Science Czech Republic (Unknown)
Responsible Party: Principal Investigator, Jan Březina, MUDr. (principal investigator), Institute for Clinical and Experimental Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F16-27449A
Record Dates: First submitted 2017-03-27; First posted 2017-04-07 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Ulcerative Colitis
Keywords: Feacal bacterial transplantation; Left-sided ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine; Enema

STUDY DESIGN:
Intervention Model Description: Patients will be split into two branches of the study by randomization criteria (gender, imunosupresive therapy). Each branch of the study will have 25-30 patients. The first group will be treated with 4 g mesalazine enema 1x daily for 2 weeks, then every other day until the end of the 6th week. A second group of patients will be applied enema prepared from 50 g of stool of examined donor dissolved in 150 ml of normal saline, the 1st week 5 times, than one time a week until the end of the 6th week.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesalazine enema (Active Comparator): Will be treated with 4 g mesalazine enema 1x daily for 2 weeks, then every other day until the end of the 6th week.
  Interventions: Drug: Mesalazine 4G Enema
- Faecal bacterial transplantation enema (Experimental): Will be applied enema prepared from 50 g of stool of examined donor dissolved in 150 ml of normal saline, the 1st week 5 times, than one time a week until the end of the 6th week.
  Interventions: Other: Faecal bacterial transplantation

INTERVENTIONS:
Other: Faecal bacterial transplantation — Enema prepared from 50 g of stool of examined donor dissolved in 150 ml of normal saline
  Other Names: FMT
  Arms: Faecal bacterial transplantation enema
Drug: Mesalazine 4G Enema — Standard mesalazine enema
  Arms: Mesalazine enema

SUMMARY:
The etiopathogenesis of ulcerative colitis (UC) is not fully understood. One of the theories of UC pathogenesis represents a pathological response of mucosal immunity to intestinal microbiota. Potential therapeutic procedure how to affect this fact is the faecal microbiota transplantation (FMT). Review of the literature on FMT suggests great potential as the treatment for UC, but two prospective controlled study that has been published yet are inconsistent.

The first objective of the project is to compare the administration of FMT enema with mesalazine enema for inducing remission in patients with active left-sided UC in the form of a prospective, randomized, controlled study. The second objective is to observe changes in the intestinal microbiota during and after FMT focusing on bacterial DNA sequencing to identify the bacterial species which are responsible for the effect of the FMT.

ELIGIBILITY:
Inclusion Criteria:

* Left-sided ulcerative colitis > 15cm ongoing more than 3 month
* Mayo score < 10
* Endoscopic Mayo score ≥ 2

Exclusion Criteria:

* Anti-TNF medication in the previous 6 months
* Cyclosporine in the previous 4 weeks
* Methotrexate in the previous 2 months
* Prednisone > 10mg
* The real risk of colectomy in the near future
* Positive stool culture (Salmonella, Shigella, Yersinia, Campylobacter, pathogenic E. coli)
* CMV infection
* Pregnancy, breastfeeding women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Clinical remission | Week 12
  Mayo score ≤ 2 with no subscore > 1

SECONDARY OUTCOMES:
Endoscopic remission | Week 6 and 12
  Mayo endoscopic score = 0
Clinical response | Week 6 and 12
  Decrease of Mayo score ≥ 2

CONTACTS AND LOCATIONS:
Locations (9):
- Czechia (9):
  - Gastroenterology departement Hospital České Budějovice, České Budějovice, Jihočeský kraj
  - Centrum péče o zažívací trakt Vítkovická nemocnice, Ostrava - Vitkovice, Moravskoslezský kraj
  - Second department of internal medicine of University Hospital Olomouc, Olomouc, Olomoucký kraj
  - IV. Department of Internal Medicine, General University Hospital in Prague, Prague, Prague 2
  - Internal departement of Thomayer Hospital, Prague, Prague 4
  - ISCARE, Prague, Prague 7
  - II. Department of Internal Medicine University Hospital Vinohrady, Prague
  - Institute of clinical and experimental medicine, Prague
  - Internal departement Hospital Na Bulovce, Prague

IPD SHARING:
Plan to Share IPD: No